CLINICAL TRIAL: NCT04920812
Title: Interest of Multi-omics (WES / RNA-Seq) Approach to Fight Against the Diagnostic Deadlock in Mitochondrial Diseases
Brief Title: MITOMICS : a Multi-OMICS Approach for the Diagnosis of Mitochondrial Diseases
Acronym: MITOMICS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-API-01; 2020-A02651-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mitochondrial diseases: annalysing with methology of multi-OMICS integration we will determined which RNA-Seq data (from muscle or fibroblasts) are the most informative for the interpretation of VUS identified by WES for patients suspected of mitochondrial myopathy.
  Interventions: Genetic: diagnosis of mitochondrial myopathy

INTERVENTIONS:
Genetic: diagnosis of mitochondrial myopathy — • Determination of the presence of specific molecular signatures at the RNA level in muscles and fibroblasts from patients

SUMMARY:
MITOMICS aims to determine which RNA-Seq results (from muscle or fibroblasts) are the most informative for the interpretation of VUS identified by WES for patients suspected of mitochondrial myopathy. Analysis of RNA-Seq and WES results will performed with a computational approach using an autoencoder-based method

DETAILED DESCRIPTION:
Mitochondrial diseases (MD) are rare, clinically and genetically extremely heterogeneous, caused by a deficit of energy production via the mitochondria. Mitochondria are dependent on 2 genomes mitochondrial DNA and nuclear DNA, and many pathogenic variants carried by these 2 genomes are responsible for mitochondrial diseases. The diagnostic strategies for MD patients have evolved significantly with the emergence of Next Generation Sequencing (NGS) also accelerating the identification of the responsible gene. However, the diagnostic yield remains limited and requires the development of new approaches. Previous studies showed that WES and RNA-Seq combination improves the diagnosis of MD, essentially by helping in the interpretation of identified VUS.

With MITOMICS project, we will included 66 patients suspected of a mitochondrial myopathy (clinical, histological or biochemical), with a negative mtDNA and WES NGS in trio. For each patient we will sequenced RNA from muscle and fibroblasts. Using a new innovative methology of multi-OMICS integration we will determined which RNA-Seq data (from muscle or fibroblasts) are the most informative for the interpretation of VUS identified by WES for patients suspected of mitochondrial myopathy. The results obtained will allow the interpretation of VUS and the identification of specific molecular signatures.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of a mitochondrial disease with muscular signs (clinical, histological or biochemical)
* Patients with negative mtDNA and WES NGS in trio
* Patients with routine muscle and skin biopsies available
* Blood samples from parents and / or relatives available for segregation studies
* Informed consent of the study signed by the patient or the legal representatives of the minor patient or under guardianship
* Patients affiliated to social security

Exclusion Criteria:

* Patients with suspected mitochondrial disease without muscle involvement
* Patients for whom the mtDNA NGS and WES have not been performed
* Patients with suspected mitochondrial disease with causal variant identified
* Refusal to sign the informed consent for the study
* Insufficient amount of frozen material or culture failure for fibroblasts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are seen in consultation by the genetic doctors of the different centers as part of the usual management of their mitochondrial disease.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
number of variations interpreted as responsible for the Mitochondrial diseases | baseline
  • Comparison of the number of variations (splicing variant, expression level) or VUS, identified in WES, interpreted as responsible for the disease (class 4 or 5 variants) thanks to the RNA-Seq carried out at from a muscle biopsy or RNA-Seq performed from fibroblasts

SECONDARY OUTCOMES:
RNA in mitochondiral deseases | baseline
  Patients for whom the RNA-Seq could not be performed and reason for failure
variation of RNA in mitochondiral deseases | baseline
  Variations identified by RNA-Seq, allowing interpretation of WES data (splicing aberrants, monoallelic expressions, etc.)
specific molecular signatures of mitochondiral deseases | baseline
  Determination of the presence of specific molecular signatures at the RNA level in muscles and fibroblasts from patients

CONTACTS AND LOCATIONS:
Overall Officials: SYLVIE BANNWARTH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (8):
- France (8):
  - CHU de Nice, Nice, CHU de NICE
  - C.H.R.U. Brest, Brest, France
  - Chu de Nantes, Nantes, France
  - chu Angers, Angers
  - Chu Brest, Brest
  - APHM, Marseille
  - Chu Montpellier, Montpellier
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No